CLINICAL TRIAL: NCT05152329
Title: Investigating the Potential Psychological Impact of Early Screening and Long-term Monitoring for Adolescent Idiopathic Scoliosis Among Patients and Caregivers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Kenny Kwan, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW19-088
Record Dates: First submitted 2021-09-28; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Adolescent Idiopathic Scoliosis; AIS; Scoliosis
Keywords: Psychological impact
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adolescent Idiopathic scoliosis (AIS) is a three-dimensional deformity of the spine of unknown aetiology, characterised by a lateral curvature and vertebral rotation. Its prevalence is estimated to be 2.5% in children between aged 10 and 16 in Hong Kong. Despite concerns regarding the psycho-social issues patients face at and after AIS screening, there is no study that directly address this subject. The investigator propose to conduct a prospective longitudinal study on the psycho-social impact of AIS early screening and long-term monitoring amongst patients and their caregivers. The proposed study will bridge this research gap by evaluating a cohort of newly-diagnosed patients with AIS through the school screening program and their caregivers. A mixed-methods research approach to tap into the distinct social, behavioural, emotional and parental experiential profiles will be used. Patterns across different profiles can enhance the investigator's understanding of which aspects of AIS early screening and long-term monitoring can adversely affect patients' psychological well-being. Findings will facilitate targeted approaches to address specific psycho-social impact of scoliosis and its treatment, heighten compliance to long-term monitoring and prevention of scoliosis progression, and mobilise a new clinical care model that addresses patient and clinician concerns.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of structural scoliosis, and
2. developmentally normal cognitive function

Exclusion Criteria:

1. A nonspinal cause of scoliosis, patients who do not intend to stay in this country for the duration of treatment, and
2. those who cannot fill in the questionnaires

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of 150 patients and their caregivers will be recruited. New referral cases to spine clinic for Adolescent Idiopathic Scoliosis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Health practices | Change from baseline health practices at 6 months
  Patients will answer questions about physical activity based on a modified version of the Paffenbarger Physical Activity Questionnaire [45], which includes questions about typical weekly energy expenditure and the duration of brisk physical activity per week. The activity score is obtained in units of kilocalorie/week, where a high value indicating high physical activity and a low value indicating low physical activity. There is no range for this scale.
General quality of life: Short-Form Health Survey (SF-12) | Change from baseline health practices at 6 months
  Generic Quality of life will be assessed through the 12-item Short-Form Health Survey (SF-12), which consists of 12 items in the physical and mental domains (Physical Component Summary (PCS)-12 and Mental Component Summary (MCS)-12; scoring range from 0-100). Higher PCS and MCS scale indicating better physical and mental health functioning.
General quality of life: European Quality of Life 5 Dimension | Change from baseline health practices at 6 months
  Generic quality of life will also be assessed through the European Quality of Life Five Dimension, which consists of five items (mobility, selfcare, usual activities, pain/discomfort and anxiety/depression). Classification scores can be linked to a utility score with 0 indicating 'death' and 1 indicating 'full health'[47].
Visual Analogue Scale | Change from baseline health practices at 6 months
  The European Quality of Life 5 Dimension (EQ-5D) is complemented by a visual analogue scale on current health, the valuation of own health, which is anchored at the lower end (0) by 'worst imaginable health state' and at the upper end (100) by 'best imaginable health state'.
Scoliosis-specific Quality of Life | Change from baseline health practices at 6 months
  Scoliosis-specific Quality of Life will be assessed through Scoliosis Research Society (SRS)-22, which consists of five domains: function/activity, pain, self-image/appearance, mental health and satisfaction with management. The SRS-22 standardises the quantification of an individual patient's views and comments in order to evaluate the results of treatment on a global basis. Each question from the SRS-22 consists of five options scored from 1 to 5. The higher the score, the more satisfied the patient is.
Body image | Change from baseline health practices at 6 months
  A modified version of the Body Image Disturbance Questionnaire (BIDQS) which specifically evaluates how scoliosis-related appearance concerns impact psychosocial and daily functioning will be used [2]. The BIDQ-S includes seven items that are scored on a scale of 1 to 5, with 5 being the highest level of body image disturbance. The overall score is calculated by obtaining the mean from all 7 questions, with score ranging from 7 to 35. A higher overall score indicating higher level of body image disturbance. In addition, the BIDQ-S includes qualitative questions inviting free text responses so that specific concerns and their impact on daily functioning can be assessed.
Parental Caregiving Experience - parental distress | Change from baseline health practices at 6 months
  Parental distress will be evaluated through the parental distress subscale of the Parenting Stress Index Short Form (PSI-SF). The subscale consisted of 12 items, rated from 1 (strongly disagree) to 5 (strongly agree), with subscales scores ranging from 12 to 60. A higher score would indicate higher level of parental distress.
Parental Caregiving Experience - Overprotection | Change from baseline health practices at 6 months
  The Overprotecting Parent Scale (VCOPS) will be used to index the degree to which the parent perceives participant's child being vulnerable and the degree to which participant display protective behaviors. VCOPS consisted of 28 items, rated from 1 "strongly agree" to 6 "strongly disagree", with score ranging from 28 to 168. A low score would indicate highly overprotective, whereas a high score would indicate an optimal level of overprotection.
Misconception | Change from baseline health practices at 6 months
  Parents will be asked to complete the True/False scale which include statements about AIS treatment options. Including this measure in the proposed study will allow us to ascertain the longitudinal predictors of continued AIS misconception(s).

CONTACTS AND LOCATIONS:
Locations (1):
- Duchess of Kent Children's Hospital, Hong Kong, Hong Kong